CLINICAL TRIAL: NCT00494819
Title: Discriminate Validity of ADHD Subtypes Using Neuropsychological Test
Brief Title: Validity of ADHD Subtypes Using Neuropsychological Measure
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9461700916; NSC 94-2815-C-002-177-H (Other: National Science Council)
Record Dates: First submitted 2007-06-29; First posted 2007-07-02 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2008-08

CONDITIONS: Attention-deficit/Hyperactivity Disorder
Keywords: ADHD, subtype, methylphenidate, neuropsychological measures
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Background: Attention-Deficit/Hyperactivity Disorder (ADHD), characterized by inattention, hyperactivity, and impulsivity, is among the most common neuropsychiatric disorders worldwide (5-10% at school age) and in Taiwan (7.5%). The DSM-IV ADHD consists of three subtypes: predominantly Inattentive (ADHD-I), predominantly Hyperactivity/Impulsivity (ADHD-H), and Combined subtypes (ADHD-C). Although the DSM-IV field trials indicate that the current subtypes differ significantly on variables such as age of onset, gender ratio, and level of social and academic impairment, little has been addressed whether the DSM-IV subtypes differ neuropsychologically. Numerous researches have proved that stimulants (methylphenidate is the only stimulant in Taiwan) are the most effective medication in treating ADHD. Although the efficacy of methylphenidate on behavioral measures has been established in Taiwan, there is no information about neuropsychological measures.

Specific Aims:

1. to validate ADHD subtype by neuropsychological measures; and
2. to investigate the efficacy of methylphenidate on the improvement of executive functioning among children with ADHD.

Subjects and Methods: Participants will consist of 20 children with ADHD-C, 20 with ADHD-I, 10 with ADHD-H and 50 controls without ADHD in the age range of 7 to 10. The measures include the psychiatric interviews (Chinese K-SADS-E), neuropsychological tests (WISC-III, Cancellation Test, Digit Span, Trail Making Test, CPT, Circle Tracing Test), self-administered rating scale (SNAP-IV), and investigator administered assessment (CGI and Behavior Observation Ratings).

Anticipated Results: We anticipated that children in the ADHD and non-ADHD group will perform differently on the neuropsychological tests with more deficits in neuropsychological functions in the ADHD group. Also, we expected that methylphenidate will improve the performance on the neuropsychological tests and reduce the behavioral symptoms of ADHD children. Subtypes difference in the neuropsychological functions is also expected.

DETAILED DESCRIPTION:
BACKGROUND AND SIGNIFICANCE Attention-Deficit/Hyperactivity Disorder (ADHD) is among the most common impairing neuropsychiatric disorder worldwide among children and adolescents with the prevalence of DSM-IV ADHD in the range of 5-10% in Western countries (Faraone et al., 2003) and 7.5% in Taiwan (Gau et al., 2005) with the ratio of boys to girls as 3-8:1. The significance of ADHD in clinical practice and research is not only in its high prevalence but also in the impairments it brings about in neurocognitive function, academic performance, and social adjustment.

The DSM-IV ADHD is comprised with three subtypes, predominantly Inattentive (ADHD-I), predominantly Hyperactivity/Impulsivity (ADHD-H), and Combined subtype (ADHD-C). The DSM-IV field trials indicate that the current subtypes differ significantly on variables such as age of onset, gender ratio, and level of social and academic impairment (Lahey et al., 1994). Although previous researches have suggested that neuropsychological deficits in ADHD are associated with frontal-subcortical regions (Castellanos, 1997), few studies have addressed whether the DSM-IV subtypes differ neuropsychologically with inconsistent results (Nigg et al, 2002).

Many studies have demonstrated the efficacy of stimulants in treating ADHD. Among them, methylphenidate (MPH) was the widely used and has been rigorously studied (eg. Spencer et al., 2005; Stein et al., 2005; Wilens et al., 2005). MPH is also the only stimulant medication for the treatment of ADHD in Taiwan; it has been proved to reduce significantly the symptoms of ADHD, and to increase self regulation, learning motivation, academic performance, and interpersonal ability. Meanwhile, its efficacy was also observed in the significant improvement of neuropsychological functioning (e.g., Konrad et al., 2004).

Given that there is no conclusive finding in the neuropsychological function among ADHD subtypes and little is known about the neuropsychological deficits in three ADHD subtypes in the Chinese population, the present study aims to validate ADHD diagnosis and ADHD subtypes by executive functioning measures. Although the efficacy of methylphenidate on behavioral measures has been established in Taiwan, there is no information about neuropsychological measures.

SPECIFIC AIMS:

1. to validate ADHD subtype by neuropsychological measures; and
2. to investigate the efficacy of methylphenidate on the improvement of executive functioning among children with ADHD.

HYPOTHESIS:

We hypothesize that ADHD and ADHD subtype can be validated by the measures of executive function and the methylphenidate not only decrease ADHD core symptoms but also improve executive functions among children with ADHD.

METHOD Participants The sample will consist of 50 child psychiatric patients with ADHD (20 ADHD-I, 20 ADHD-C and 10 ADHD-H) and 50 normal controls, aged 7-10. The inclusion criteria are patients who have clinically diagnosis of DSM-IV ADHD confirmed by the K-SADS-E, are aged 7-10, and have IQ > 80; and who and whose parents consent to this study. Participants will be excluded if they have a history of brain injury or epilepsy, visual/auditory deficit or were diagnosed as having motor disorder, obsessive-compulsive disorder, mental retardation, and depression. In order to recruit a population of pure ADHD (without other psychiatric comorbidities), children who are comorbid with oppositional defiant disorder (ODD) or conduct disorder (CD) were excluded, though the concurrence of ODD/CD and ADHD were high. Normal controls will be recruited from the local elementary school in the same geographical area.

Measurements Considering the age group selected and symptoms of ADHD, we selected measurements carefully to ensure that all participants will be able to complete every task without getting fatigued or being distractive in the task.

1. Chinese version of the Kiddie-Schedule for Affective Disorders and Schizophrenia- epidemiology version (K-SADS-E) Development of the Chinese K-SADS-E was carried out by the Child Psychiatry Research Group in Taiwan, which included a two-stage translation and modification of several items with psycholinguistic equivalents relevant to the Taiwanese culture. The K-SADS-E has been widely used in a variety of studies on the mental illness of children and adolescents in Taiwan (Gau et al., 2005). Mother will be interviewed independently by two separate interviewers to make child's psychiatric diagnoses.
2. Wechsler Intelligence Scale for Children Short Form (WISC-III short form) WISC-III (Wechsler, 1991) is a well established scale designed to assess the Full-Scale IQ (FSIQ) of children under age of 16. It includes 13 subtests to test children's cognitive ability of different dimensions. Test result is represented by Verbal IQ, Performance IQ, and Full-Scale IQ. The present research conducted a quad combination of WISC short form including subtests of Symbol Search, Arithmetic, Block Design, and Verbal. Previous research suggested the mentioned combination have good reliability (rxx = .91) and validity (rxx = .90) (Silverstein, 1982), and is preferred while conducting research to estimate FSIQ.
3. Neuropsychological measures Five neuropsychological measures which consist of 19 task variables will be used.

   Cancellation Test (Rudel et al., 1978) Cancellation Test is a two-part paper-and-pencil measure of visual scanning. Number Cancellation requires subject to strike out a three-digit target (257) intermittently placed in a large array of numbers; Shape Cancellation required subject to strike out a target shape (star) intermittently place in a filed of other shapes. The total number of commission error, correct hits, and completed time on the two separate tests will be recorded. Completion time divided by the number is calculated as one of the indices.

   Digit Span The assessor first requires subjects to repeat orally presented digit strings (Digit Forward) and then recall digits in backwards sequence (Digit Backward). This task represents the indices of sensory selection and capacity/focus components, in the present research.

   Trail Making Test (TMT; Reitan & Wolfson, 1986) A brief paper-and-pencil test involving numeric sequencing (Trail A) followed by alpha-numeric sequencing (Trail B) in original form. The Trail B was modified by using Chinese phonic symbols to substitute for English alphabet when applying to Chinese participants. Completed time and off-target errors on the tasks are oriented to the attentional components of sensory selection, response selection, and capacity/focus.

   Continuous Performance Test (CPT; Conners, 1995) The CPT requires tabbing on the space key when any character other than X shown on the screen. There were six sets in total, with 20 characters within each set. The Inter-Stimulus Intervals (ISIs) are 1, 2, and 4 seconds, and different ISIs varied between sets. Each character maintains on the screen for 250 ms. Correct hits, omission errors, commission errors, and reaction times will be collected as indices of response selection and capacity/focus. The d' value known as a discriminate factor is one of the indices for sustained attention.

   Circle Tracing Test (CTT, Bachorowski & Newman, 1985) This task requires subjects to trace a large printed circle (20 inches in diameter) with their index finger to measure inhibition of an ongoing response (eg. Geurts et al, 2004; Scheres et al., 2003). The word START (in green ink) was printed on the right side of the line and the word STOP (in red ink) was printed on the left side. The task was administered under two conditions: first with neutral instruction ('trace the circle') followed by inhibition instruction ('trace the circle again, but as slow as you can this time') within 12 minutes without subject's knowledge. The dependent variable on this task included time 1 under neutral instruction, time 2 under inhibition instruction, time discrepancy referred to time 2 minus time 1, and a three-point (0-2) degree of deviation score assessed by the trained observer. The larger the time discrepancy, the better a participant is able to inhibit (slow down) the continuous tracing response.
4. Measures of behavior symptoms Subjects' parent will complete the SNAP-IV and a trained rater will observe the subjects' behaviors and rate on two behavioral scales during the tasks.

Swanson, Nolan, and Pelham IV scale (SNAP-IV, Swanson et al., 2001) The SNAP-IV is a 26-item rating scale consisting of the DSM-IV symptoms for the Inattention (Item 1-9) and the Hyperactivity/Impulsivity domains (Item 10-18) of the criteria for ADHD, and the oppositional symptoms (Item 19-26) of the criteria for ODD. Several studies have used different versions of the SNAP, either parent or teacher form, as an outcome measure to assess the efficacy of treatment for ADHD (e.g., Steele et al., 2006). Regarding psychometric properties of the SNAP rating scale, the Chinese version of SNAP-IV showed satisfactory test-retest reliability (intraclass correlation= 0.59~0.72), internal consistency (alpha=0.88~0.90), concurrent validity (Pearson correlations = 0.56~0.72), and discriminant validity (Liu et al., 2006).

Clinical Global Impression (CGI, NIMH, 1976) CGI, a three-item scale including Severity of Illness, Global Improvement, and Efficacy Index, is used to assess treatment response in psychiatric patients. The Severity of Illness with 7-point scale (1 = normal to 7 = extremely ill) will be used in this study.

Behavior Observation Ratings This is a four-point (0 = not at all to 3 = extremely much) rating scales with three items assessing children's behaviors during the task. The three target behaviors to be observed are "unsteady while remaining seated," "murmuring during task," and "given up easily" before and after one dose of methylphenidate.

Procedure We will obtain written informed consent of all subjects from both children and their parents. The day prior to the date of receiving neuropsychological tasks, children will be asked to halt medication in order to obtain their test results as baseline data to make comparison with their performance after treatment with MPH.

The testing procedure is as follows: (1) All children (ADHD group and normal controls) will be assessed IQ and a series of neuropsychological assessments. Their parents will complete the SNAP-IV scale at the same time. (2) After that, children with ADHD will take IR MPH (at the same dose as their prescription) and rest for approximately 45 minutes. Meanwhile, parents of children with ADHD will be interviewed with K-SADS-E by trained interviewer. (3) Children with ADHD will then be re-assessed CPT. CGI and Behavior observation will be assessed.

ANTICIPATED RESULT We anticipated that children in the ADHD and non-ADHD group will perform differently on the neuropsychological tests with more deficits in neuropsychological functions in the ADHD group. Also, we expected that methylphenidate will improve the performance on the neuropsychological tests and reduce the behavioral symptoms of ADHD children. Subtypes difference in the neuropsychological functions is also expected.

CONCLUSION The present research aims to inspect the effect of methylphenidate on behavioral measures and neuropsychological function among children with ADHD in Taiwan. Understanding the treatment effect among neuropsychological function and different behavior may help us clear out the psychopathology of ADHD. Learning the possible difference among subtypes regarding the relationship of treatment and self-report outcome will benefit in that matter as well.

ELIGIBILITY:
Inclusion Criteria:

* patients who have clinically diagnosis of DSM-IV ADHD confirmed by the K-SADS-E, are aged 7-10, and have IQ > 80; and who and whose parents consent to this study

Exclusion Criteria:

* if they have a history of brain injury or epilepsy, visual/auditory deficit or were diagnosed as having motor disorder, obsessive-compulsive disorder, mental retardation, mood disorders, pervasive developmental disorder, or schizophrenia

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 122 (Actual)
Dates: Start 2005-09; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiang M, Gau SS. Validation of attention-deficit-hyperactivity disorder subtypes among Taiwanese children using neuropsychological functioning. Aust N Z J Psychiatry. 2008 Jun;42(6):526-35. doi: 10.1080/00048670802050603. PMID 18465380